CLINICAL TRIAL: NCT04904159
Title: A New Scoring System in the Diagnosis of Thyroid Gland Pathologies
Brief Title: Scoring System for Thyroid Gland Pathologies
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ramazan Sari, Principal Investigator, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: 2021/514/198/20
Record Dates: First submitted 2021-05-17; First posted 2021-05-27 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Thyroid Nodule; Thyroid Cancer
Keywords: TI-RADS; Bethesda
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms | interventions — Thyroidectomy; Anterior Temporal Lobectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Benign: Patients who have benign pathologies after thyroidectomy
  Interventions: Procedure: Lobectomy
- Malign: Patients who have malign pathologies after thyroidectomy
  Interventions: Procedure: Thyroidectomy

INTERVENTIONS:
Procedure: Thyroidectomy — total thyroidectomy
  Groups: Malign
Procedure: Lobectomy — Lobectomy
  Groups: Benign

SUMMARY:
Although anamnesis and physical examination remain the place in the evaluation of patients today; laboratory values, imaging methods and pathology results have come to the fore in the decision-making of surgery for patients. As a result of all other criteria, a follow-up decision can be changed in a patient with a single fine needle aspiration biopsy result, or despite all the examinations the investigators have, a clear result cannot be achieved, and patient management may be disrupted. A holistic approach to thyroid gland pathologies is planned thanks to the scoring system that will be created in this study.

DETAILED DESCRIPTION:
In routine clinical practice, the criteria the investigators consider during the pre - op period in patients evaluated due to thyroid pathologies include anamnesis, physical examination, laboratory values, especially thyroid function, thyroid-neck ultrasonographies, fine needle aspiration biopsies, according to which decisions about operation or nonoperative follow-up are made with the patient. The investigators aim to create a common scoring system by taking into account the pathology results of patients who have undergone thyroidectomy and comparing these results with the results of pre-op examination and thus to address patient management in a more objective and comprehensive way.

ELIGIBILITY:
Inclusion Criteria:

* patients who undergone surgery for thyroid gland pathologies

Exclusion Criteria:

* patients who did not want to be involved in the study
* patients who missed in the follow-up period
* pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thyroidectomy, which is a routine operation in clinic ( unilateral, total, complementary, etc.) ) applied patients will be included in the study
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Age | Before Surgery
  Years
Gender | Before Surgery
  Male - Female
Smoking Status | Before Surgery
  Yes or No
Radiation to the Neck Area | Before Surgery
  Yes or No
History of Thyroiditis | Before Surgery
  Yes or No
Family History | Before Surgery
  Presence of family members with any thyroid pathologies especially thyroid cancer
Complaint | Before Surgery
  Months
Thyroid Imaging Reporting and Data System ( TIRADS ) score | Before surgery
  Radiological features of throid nodule ( minimum value is 1 maximum value is 5 ); thyroid nodule which has a higher value means a worse outcome
Bethesda classification system for thyroid fine needle aspirates | Before surgery
  Histopathological features of thyroid nodule ( minimum value is 1 maximum value is 6 ) thyroid nodule which has higher value means a worse outcome
Thyroid Stimulating Hormone ( TSH ) levels | Before surgery
  it is a hormone secreted from the pituitary gland and triggers the functioning of the thyroid gland ( cut of values are 0.5 - 5.0 mIU / L )
Pathology results | Immediately after the surgery
  The result of the throid gland part sent to the pathology unit after surgery ( the results can be benign or malign )

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Fehmi Küçük, Prof., Study Chair — Istanbul Dr. Lutfi Kirdar Kartal Training and Research Hospital
Locations (1):
- Kartal Dr Lutfi Kirdar Tranining and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macias CA, Arumugam D, Arlow RL, Eng OS, Lu SE, Javidian P, Davidov T, Trooskin SZ. A risk model to determine surgical treatment in patients with thyroid nodules with indeterminate cytology. Ann Surg Oncol. 2015 May;22(5):1527-32. doi: 10.1245/s10434-014-4190-8. Epub 2014 Nov 12. PMID 25388058
- [Background] Ianni F, Pascucci D, Paragliola RM, Rota CA, Perotti G, Fadda G, Pontecorvi A, Corsello SM. Follow-Up or Surgery for Indeterminate Thyroid Nodules: Could the CUT Score Application Be a Support for Decision-Making in the Preoperative Assessment? Thyroid. 2020 Jan;30(1):65-71. doi: 10.1089/thy.2018.0649. Epub 2019 Oct 23. PMID 31552809
- [Background] Sparano C, Verdiani V, Pupilli C, Perigli G, Badii B, Vezzosi V, Mannucci E, Maggi M, Petrone L. Choosing the best algorithm among five thyroid nodule ultrasound scores: from performance to cytology sparing-a single-center retrospective study in a large cohort. Eur Radiol. 2021 Aug;31(8):5689-5698. doi: 10.1007/s00330-021-07703-5. Epub 2021 Feb 18. PMID 33599836
- [Background] Shin HS, Na DG, Paik W, Yoon SJ, Gwon HY, Noh BJ, Kim WJ. Malignancy Risk Stratification of Thyroid Nodules with Macrocalcification and Rim Calcification Based on Ultrasound Patterns. Korean J Radiol. 2021 Apr;22(4):663-671. doi: 10.3348/kjr.2020.0381. Epub 2021 Feb 2. PMID 33660454
- [Background] Madeo B, Brigante G, Ansaloni A, Taliani E, Kaleci S, Monzani ML, Simoni M, Rochira V. The Added Value of Operator's Judgement in Thyroid Nodule Ultrasound Classification Arising From Histologically Based Comparison of Different Risk Stratification Systems. Front Endocrinol (Lausanne). 2020 Jul 7;11:434. doi: 10.3389/fendo.2020.00434. eCollection 2020. PMID 32733383
- [Background] Cozzolino A, Pozza C, Pofi R, Sbardella E, Faggiano A, Isidori AM, Giannetta E, Pernazza A, Rullo E, Ascoli V, Lenzi A, Gianfrilli D. Predictors of malignancy in high-risk indeterminate (TIR3B) cytopathology thyroid nodules. J Endocrinol Invest. 2020 Aug;43(8):1115-1123. doi: 10.1007/s40618-020-01200-0. Epub 2020 Feb 25. PMID 32100197
- [Background] Maia FF, Matos PS, Pavin EJ, Zantut-Wittmann DE. Thyroid imaging reporting and data system score combined with Bethesda system for malignancy risk stratification in thyroid nodules with indeterminate results on cytology. Clin Endocrinol (Oxf). 2015 Mar;82(3):439-44. doi: 10.1111/cen.12525. Epub 2014 Jul 7. PMID 24930423
- [Background] Remonti LR, Kramer CK, Leitao CB, Pinto LC, Gross JL. Thyroid ultrasound features and risk of carcinoma: a systematic review and meta-analysis of observational studies. Thyroid. 2015 May;25(5):538-50. doi: 10.1089/thy.2014.0353. Epub 2015 Mar 31. PMID 25747526
- [Background] Chaigneau E, Russ G, Royer B, Bigorgne C, Bienvenu-Perrard M, Rouxel A, Leenhardt L, Belin L, Buffet C. TIRADS score is of limited clinical value for risk stratification of indeterminate cytological results. Eur J Endocrinol. 2018 Jul;179(1):13-20. doi: 10.1530/EJE-18-0078. Epub 2018 Apr 27. PMID 29703794